CLINICAL TRIAL: NCT04712955
Title: Bloodflow Restricted Exercise in Healthy Ageing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 190824010610
Record Dates: First submitted 2021-01-08; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Aging
Keywords: bloodflow restricted exercise; skeletal muscle; muscle stem cells

STUDY DESIGN:
Intervention Model Description: Single center randomised controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bloodflow restricted exercise (Active Comparator): Healthy subjects undergoing low intensity blood flow restricted resistance exercise (BFRRE) conducted as 4 sets of bilateral knee extensions at 30% of 1RM until voluntary fatigue. The sets are intercepted by 30 seconds of rest (during rest the cuff's are still inflated).
  Interventions: Other: Bloodflow restricted exercise
- Non-exercise control (No Intervention): No intervention.

INTERVENTIONS:
Other: Bloodflow restricted exercise — Low-intensity bloodflow restricted resistance exercise is conducted as traditional knee extension exercise with a load corresponding to 30% of 1 repetition maximum (RM), with concurrent partial occlusion of the circulation by means of inflatable pneumatic cuffs wrapped around the proximal part of the thighs. Cuffs are inflated to a pressure corresponding to 50% of the arterial occlusion pressure, which only compromises venous but not arterial blood flow.
  Other Names: BFRRE
  Arms: Bloodflow restricted exercise

SUMMARY:
The overall objective of this study is to investigate the efficacy of low-intensity blood flow restricted resistance exercise (BFRRE) to promote health beneficial skeletal muscle adaptations and augment muscle function in a healthy older population. This objective will be achieved by in-dept evaluation of skeletal muscle cellular and functional characteristics prior to and after an intervention period comprising 6 weeks of BFRRE or non-exercise control intervention in healthy older subjects. A special focus is placed on the ability of BFRRE to stimulate skeletal muscle protein synthesis and augment muscle stem cell function.

Furthermore, recent findings suggests that similar exercise interventions in a population of patients with heart failure (HF) does not stimulate the desired adaptations. In accordance, we aim to compare the adaptive response to BFRRE amongst HF patients and the enrolled age-matched healthy individuals from the present investigation.

The findings of the current study will expand our understanding of how low-intensity resistance exercise alternatives might be viable in promoting muscle anabolism to combat the loss of muscle mass observed with ageing as well as the potential anabolic resistance accompanying HF diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the written and spoken information and to give informed consent for inclusion.
* Age between 45 and 80 years
* Able to sit in a knee extension machine
* Able to deliver muscle biopsies
* Able to train 3 times per week during a 6-week period

Exclusion Criteria:

* Known history of cardiac disease
* Habitual exercise with high intensity > 2 times pr. week within the past 6 months
* Pregnancy
* Diabetes mellitus
* Peripheral neuropathy
* Dialysis treatment
* Severe peripheral arterial disease
* Concomitant acute life threatening medical condition
* Intracranial aneurisms, arteriovenous malformation, cerebral neoplasm or abscess
* Severe arterial hypertension (≥ 180/≥ 110 mmHg) or moderate arterial hypertension (160-179/100-109) despite medical treatment
* Moderate or severe chronic obstructive pulmonary disease
* Decreased kidney function - eGFR < 60 ml/min

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-19 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Subfractional muscle protein synthesis rates | 6 weeks
  Myofibrillar protein synthesis rate
Subfractional muscle protein synthesis rates | 6 weeks
  Mitochondrial protein synthesis rate
Segmental muscle mass of lower extremity | 6 weeks
  Dual Energi X-ray Absorption (DEXA)
Muscle fibre cross sectional area (CSA) | 6 weeks
  Histological examination of muscle biopsies
Muscle stem cell function | 6 weeks
  Time to first division
Muscle stem cell function | 6 weeks
  Proliferative capacity
Muscle stem cell function | 6 weeks
  Differentiation capacity

SECONDARY OUTCOMES:
Maximal Voluntary Contraction (MVC) | 6 weeks
  Isometric muscle function
1 repetition maximum | 6 weeks
  Dynamic muscle strength
Muscle strength-endurance capacity | 6 weeks
  Local muscle endurance

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Vissing, PhD, Study Director — University of Aarhus
Locations (1):
- University of Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Groennebaek T, Jespersen NR, Jakobsgaard JE, Sieljacks P, Wang J, Rindom E, Musci RV, Botker HE, Hamilton KL, Miller BF, de Paoli FV, Vissing K. Skeletal Muscle Mitochondrial Protein Synthesis and Respiration Increase With Low-Load Blood Flow Restricted as Well as High-Load Resistance Training. Front Physiol. 2018 Dec 17;9:1796. doi: 10.3389/fphys.2018.01796. eCollection 2018. PMID 30618808
- [Background] Sieljacks P, Wang J, Groennebaek T, Rindom E, Jakobsgaard JE, Herskind J, Gravholt A, Moller AB, Musci RV, de Paoli FV, Hamilton KL, Miller BF, Vissing K. Six Weeks of Low-Load Blood Flow Restricted and High-Load Resistance Exercise Training Produce Similar Increases in Cumulative Myofibrillar Protein Synthesis and Ribosomal Biogenesis in Healthy Males. Front Physiol. 2019 May 29;10:649. doi: 10.3389/fphys.2019.00649. eCollection 2019. PMID 31191347
- [Background] Groennebaek T, Sieljacks P, Nielsen R, Pryds K, Jespersen NR, Wang J, Carlsen CR, Schmidt MR, de Paoli FV, Miller BF, Vissing K, Botker HE. Effect of Blood Flow Restricted Resistance Exercise and Remote Ischemic Conditioning on Functional Capacity and Myocellular Adaptations in Patients With Heart Failure. Circ Heart Fail. 2019 Dec;12(12):e006427. doi: 10.1161/CIRCHEARTFAILURE.119.006427. Epub 2019 Dec 13. PMID 31830830